CLINICAL TRIAL: NCT06733324
Title: Randomized Control Trial of SCERTS (Social Communication, Emotional Regulation, Transactional Support) Program for Children With Autism Spectrum Disorder
Brief Title: RCT of SCERTS (Social Communication, Emotional Regulation, Transactional Support) Program for Children With Autism Spectrum Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aisha Saleem (Other)
Collaborators: Ayub Medical College, Abbottabad (Other)
Responsible Party: Sponsor-Investigator, Aisha Saleem, Clinical Psychologist & Lecturer, National University of Science and Technology, Pakistan
Organization: National University of Science and Technology, Pakistan (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC-EA-2024/265
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Autism Spectrum Disorder (ASD
Keywords: Autism Spectrum Disorder; SCERTS; Parental Distress; Quality of Life; Adaptive Behavior
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Behavior Therapy; Speech Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participants will receive SCERTS intervention (Experimental): Participants in the experimental group will receive the SCERTS (Social Communication, Emotional Regulation, and Transactional Support) intervention program. This is an evidence-based, individualized program designed to improve social communication, emotional regulation, and adaptive behaviors in children with Autism Spectrum Disorder (ASD) aged 3-6 years. The intervention will be delivered over 8 weeks, with weekly structured sessions involving parents and educators to ensure skill generalization across home and school settings. The program includes strategies to enhance joint attention, emotion sharing, symbolic play, and the use of non-verbal cues. Parents will be actively engaged to facilitate ongoing support and reinforcement in real-life environments.
  Interventions: Behavioral: SCERTS (Social Communication, Emotional Regulation, Transactional Support)
- Control Group (Active Comparator): Participants in the treatment-as-usual (TAU) group will receive the standard care typically available for children with Autism Spectrum Disorder (ASD) in the community. This may include therapies such as speech-language therapy, occupational therapy, and applied behavior analysis, depending on the availability of services and individual needs. These interventions focus on addressing core ASD symptoms like communication deficits, behavioral challenges, and sensory integration difficulties. The TAU group will not receive any components of the SCERTS intervention during the study period. This group will serve as an active comparator to evaluate the relative effectiveness of the SCERTS program in improving social communication, emotional regulation, and adaptive behaviors. After the study concludes, participants in the TAU group will have the opportunity to receive the SCERTS intervention to ensure equitable access to the experimental treatment.
  Interventions: Behavioral: Behavioral Treatment, Speech Therapy

INTERVENTIONS:
Behavioral: SCERTS (Social Communication, Emotional Regulation, Transactional Support) — The SCERTS (Social Communication, Emotional Regulation, and Transactional Support) intervention is a comprehensive, multidisciplinary approach specifically tailored to address the unique needs of children with Autism Spectrum Disorder (ASD) aged 3-6 years. Unlike traditional behavioral therapies such as Applied Behavior Analysis (ABA), SCERTS emphasizes a developmental framework, focusing on enhancing social communication, emotional regulation, and environmental support. It incorporates family involvement and integrates strategies into naturalistic settings, ensuring skill generalization across home, school, and community environments.
  This intervention is distinguished by its individualized goals based on each child's developmental profile and its emphasis on fostering meaningful interactions rather than relying on compliance-based methods. SCERTS also incorporates transactional supports, such as modifying the physical and social environment to promote engagement and reduce stress, w
  Arms: Participants will receive SCERTS intervention
Behavioral: Behavioral Treatment, Speech Therapy — The control group will be the treatment as usual group receiving conventional behavior therapy and speech therapy
  Arms: Control Group

SUMMARY:
This randomized control trial aims to assess the efficacy of the SCERTS intervention in children aged 3-6 years diagnosed with mild to moderate Autism Spectrum Disorder (ASD). The study evaluates the program's impact on improving social communication skills, adaptive behavior, and reducing caregiver stress while enhancing parental quality of life. The intervention incorporates components of Social Communication, Emotional Regulation, and Transactional Support, tailored to cultural and contextual needs in Pakistan. The study will also validate translated and culturally adapted tools for program evaluation.

The SCERTS model is a multidisciplinary, evidence-based intervention that focuses on enhancing social communication, emotional regulation, and providing transactional support in children with ASD. This 8-week program will be tested through a single-blind randomized trial, with participants assigned to an experimental group or a waitlist control group. Outcomes include joint attention, imitation, emotional sharing, and intentional communication. The study will also evaluate the intervention's feasibility, fidelity, and acceptability in the Pakistani context. Post-intervention assessments and follow-ups will determine long-term benefits.

DETAILED DESCRIPTION:
This study is a single-blind, randomized controlled trial to evaluate the efficacy of the SCERTS (Social Communication, Emotional Regulation, Transactional Support) intervention for children with Autism Spectrum Disorder (ASD) aged 3 to 6 years. ASD is a neurodevelopmental disorder with increasing prevalence worldwide and in Pakistan, where it remains underdiagnosed and underserved. This study aims to address gaps in autism care by culturally adapting and implementing the SCERTS model in a resource-constrained setting.

The SCERTS intervention focuses on three core components: improving Social Communication (e.g., joint attention, reciprocal interaction), enhancing Emotional Regulation (e.g., coping with stress, self-regulation), and fostering Transactional Support (e.g., creating supportive environments through caregiver involvement). This family-centered approach empowers parents and teachers to implement strategies in natural settings, reducing caregiver stress while promoting child development.

The trial will enroll 30 participants, divided into an experimental group receiving the SCERTS intervention and a waitlist control group receiving standard care. The intervention spans 8 weeks, with weekly sessions involving individualized and group activities tailored to the child's developmental level and cultural context. Outcome measures include social communication skills, adaptive behaviors, caregiver stress, and quality of life, assessed using validated, culturally adapted tools.

This trial adheres to the Medical Research Council Framework for complex interventions and follows CONSORT guidelines for feasibility studies. The findings are expected to provide evidence for the effectiveness and scalability of the SCERTS model in low-resource settings, contributing to improved care and outcomes for children with ASD and their families in Pakistan.

This description is clear, comprehensive, and aligns with ClinicalTrials.gov requirements. It highlights the purpose, design, methodology, and expected significance of the study.

The main objectives of the study are:

1. To translate and validate the outcome measures for the evaluation of the program.
2. To determine the fidelity, feasibility and acceptability of implementing the SCERTS intervention in Pakistani culture, including participant recruitment, intervention delivery, and adherence to the intervention protocol.
3. To translate and culturally adapt the SCERTS Intervention Program and establish its cultural equivalence to make it suitable for Pakistani culture.
4. To assess the efficacy of the Social Communication, Emotional Regulation, and Transactional Support (SCERTS) intervention compared to standard care in improving social communication skills among children diagnosed with Autism Spectrum Disorder (ASD) aged between 3 to 6 years.
5. To investigate the effectiveness of the SCERTS intervention in promoting adaptive behaviors and functional outcomes in children with ASD aged between 3 to 6 years, as measured by standardized assessment tools.
6. To assess the maintenance of intervention effects over time through follow-up assessments conducted at specified intervals post-intervention.

The hypotheses of the study are:

1. Children with ASD who receive the SCERTS Intervention will demonstrate significant improvement in social communication skills as compared to treatment as usual group.
2. Children with ASD who receive the SCERTS program will demonstrate significant improvement in adaptive behavior as compared to TAU Group.
3. Parents and caregivers of children with ASD who participate in SCERTS intervention will report significantly higher quality of life as compared to TAU Group.
4. Parents and caregivers of children with ASD who participated in SCERTS intervention will demonstrate significant reduction in caregiver stress as compared to TAU group.

ELIGIBILITY:
Inclusion Criteria:

* Age-3 to 6 years
* Diagnosis- Mild and Moderate ASD (Based on the score of Childhood Autism Rating Scale)

Exclusion Criteria:

* Age less than 3 or more than 6
* Diagnosis: Severe Autism Spectrum Disorder, Any other neurodevelopmental disorder

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
SCERTS Assessment Process | 3 months
  Social Communication, Emotional Regulation and Transactional Support

SECONDARY OUTCOMES:
Developmental Disorders-Children Disability Assessment Schedule (DD-CDAS) | 3 to 4 months
  Addresses various domains of adaptive behavior skills
WHO Quality of Life Scale | 3 months
  To assess the overall quality of life of the family
Perceived Stress Scale | 3 months
  To measure to level of stress in primary caregivers

CONTACTS AND LOCATIONS:
Locations (1):
- Ayub Medical College and Teaching Hospital, Abbottabad, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No
Keeping in view the confidentiality